CLINICAL TRIAL: NCT03136029
Title: Overcoming Exercise Intolerance in Veterans With Heart Failure: The Role of NO
Brief Title: Exercise and NO in HFrEF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: F1311-R
Record Dates: First submitted 2017-04-27; First posted 2017-05-02 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF; Exercise Intolerance; Nitric Oxide
MeSH Terms: interventions — Antioxidants; sapropterin; Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Oral AOx (Experimental): 8 week oral antioxidant treatment
  Interventions: Dietary Supplement: Antioxidant
- Oral AOx (placebo) (Placebo Comparator): Placebo for arm 1
  Interventions: Dietary Supplement: Antioxidant
- Oral BH4 (Experimental): 8 week oral tetrahydrobiopterin treatment
  Interventions: Dietary Supplement: Tetrahydrobiopterin (BH4)
- Oral BH4 (placebo) (Placebo Comparator): Placebo for arm 3
  Interventions: Dietary Supplement: Tetrahydrobiopterin (BH4)
- Ex training (Experimental): 8-week knee-extensor exercise training program
  Interventions: Other: Exercise training
- Ex training (attn con) (Sham Comparator): Attention control for arm 5
  Interventions: Other: Exercise training

INTERVENTIONS:
Dietary Supplement: Antioxidant — Daily consumption of over-the-counter vitamins (600mg alpha lipoic acid, 1000mg vitamin c, 600IU vitamin E)
  Arms: Oral AOx; Oral AOx (placebo)
Dietary Supplement: Tetrahydrobiopterin (BH4) — Daily consumption of BH4 (10mg/kg)
  Other Names: Kuvan
  Arms: Oral BH4; Oral BH4 (placebo)
Other: Exercise training — Aerobic exercise training program (3x/week for 8 weeks, 1 hour per session)
  Arms: Ex training; Ex training (attn con)

SUMMARY:
Heart disease is the leading cause of death in the United States, accounting for one in every four deaths in 2010 and costing over $300 billion annually in health care, medication, and lost productivity. Heart failure with a reduced ejection fraction (HFrEF), a clinical syndrome that develops as a consequence of heart disease, now affects almost 6 million Americans. Within the VA Health Care System, HFrEF hospital admission rates continue to rise, and remain the number one reason for discharge from VA hospitals nationwide. Unfortunately, over one-third of all Veterans suffering from HFrEF die within two years of discharge despite optimized drug therapy, an unacceptably high number. This proposal is focused on how impaired muscle blood flow contributes to exercise intolerance in HFrEF, and on subsequently developing strategies for restoring exercise tolerance and slowing disease progression in this patient group. It is anticipated that knowledge gained from these studies will contribute to improved standard of care, quality of life, and prognosis in this VA patient group.

DETAILED DESCRIPTION:
Heart failure with reduced ejection fraction (HFrEF), a clinical syndrome that develops as a consequence of heart disease from multiple etiologies, now affects almost six million Americans, presenting an imminent need for further research addressing the pathophysiology of this pervasive disease. One of the most damaging consequences of the disease is an elevation in sympathetic nervous system (SNS) activity, which manifests peripherally as chronic vasoconstriction. In HFrEF patients, peripheral vasoconstriction acts to limit blood flow in the exercising muscle, promoting exercise intolerance, premature skeletal muscle fatigue, inactivity, and a subsequent acceleration in disease progression. Fortunately, disease-related sympathoexcitation may be remediable. Among the most influential modulators of peripheral SNS expression is the nitric oxide (NO) pathway. Thus, interventions focused on improving NO bioavailability may offer a new, unexplored strategy for inhibiting SNS overactivity in HFrEF, and thus represent a novel approach for improving and exercise tolerance.

Specific Aim 1 will utilize an oral antioxidant (AOx) cocktail to study whether disruptions in oxidative stress can favorably influence exercise tolerance in HFrEF patients.

Specific Aim 2 will examine the efficacy of oral tetrahydrobiopterin (BH4), a cofactor for endothelial nitric oxide synthase (eNOS), to improve exercise intolerance in HFrEF patients.

Specific Aim 3 will examine the therapeutic potential of aerobic, knee-extensor (KE) exercise training to improve skeletal muscle blood flow and thus exercise tolerance in HF patients. Importantly, this exercise modality produces a potent training stimulus without the significant cardiopulmonary stress that accompanies more traditional, whole-body exercise. It is proposed that 12 weeks of supervised KE training will increase NO bioavailability and inhibit SNS activity, which will in turn improve vascular function and exercising limb blood flow.

Specific Aim 4 will examine whether the interventional strategies in Aims 1-3 can improve adherence to an 8-week clinical cardiac rehabilitation program. It is hypothesized that chronic AOx consumption (Aim 1), BH4 consumption (Aim 2), and aerobic exercise training (Aim 3) interventions will reduce the rate of attrition from Phase II outpatient Cardiac Rehabilitation in HFrEF patients compared to patients that did not participate in an interventional phase of the study.

The investigators anticipate that disrupting this "vicious cycle" of vasoconstriction in HFrEF may improve overall vascular health to such a degree that significant improvements in exercise-related symptoms are realized, which could therefore improve enrollment in a cardiac rehabilitation program. In this context, findings from the proposed work may provide an important link between vascular and rehabilitative medicine, thus serving to refine current strategies for the treatment of Veterans with HFrEF, ultimately leading to enhanced quality of life in this cohort.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion/Exclusion Criteria:

* The study group will include subjects with a history of stable cardiomyopathy (ischemic and non-ischemic, >3 months duration, ages 45-75 yrs) despite a minimum of 6 weeks of optimal treatment.
* Optimal therapy will be according to American Heart Association (AHA) /American College of Cardiology (ACC) and Heart Failure Society of America (HFSA) HF guidelines, including treatment with angiotensin-converting enzyme (ACE) and -blocker therapy (for at least 6 weeks), or have documented reason for variation, including medication intolerance, contraindication, patient preference, or personal physician's judgment.
* Patient enrollment will be limited to those individuals with New York Heart Association (NYHA) class II and III symptoms, left ventricular ejection fraction <35% (LVEF), with no or minimal smoking history (<15 pk yrs), and without pacemakers.

Exclusion Criteria:

* Patients with atrial fibrillation or HF believed to be secondary to atrial fibrillation will be excluded.
* Patients with HF secondary to significant uncorrected primary valvular disease (except mitral regurgitation secondary to left ventricular dysfunction) will also be excluded.
* Patients will be sedentary, defined here as no regular physical activity for at least the prior 6 months and current activity level will be documented by an activity questionnaire.
* Patients must have no orthopedic limitations that would prohibit them from performing knee-extensor exercise.
* Due to the typical age of patients with HF, all women will be postmenopausal (either natural or surgical) defined as a cessation of menses for at least 2 years, and in women without a uterus, follicle stimulating hormone (FSH) >40 IU/L.
* Women currently taking hormone replacement therapy (HRT) will be excluded from the proposed studies due to the direct vascular effects of HRT Comorbidity Exclusion Criteria: Patients with significant non-cardiac comorbidities, which if present could alter the study results, will be excluded.

  * These include a diagnosis of Dementia
  * Severe chronic obstructive pulmonary disease (COPD)
  * Peripheral Vascular Disease
  * Anemia
  * Sleep-related Breathing Disorder
  * Severe Valvular Heart Disease
  * Diabetes (if on insulin therapy)
  * or End-stage Malignancy
* The investigators will also exclude morbidly obese patients (BMI >40), patients with uncontrolled Hypertension (>160/100), Anemia (Hgb<9) and Severe Renal Insufficiency (individuals with creatinine clearance <30 by the Cockcroft-Gault formula).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Blood Flow | four years
  ultrasound Doppler

CONTACTS AND LOCATIONS:
Overall Officials: David W. Wray, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No